CLINICAL TRIAL: NCT04925479
Title: A Multi-center, Open-label Study to Determine the Dose and Safety of Oral Asciminib in Pediatric Patients With Philadelphia Chromosome Positive Chronic Myeloid Leukemia in Chronic Phase (Ph+ CML-CP), Previously Treated With One or More Tyrosine Kinase Inhibitors
Brief Title: Study to Determine the Dose and Safety of Asciminib in Pediatric Patients With Chronic Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CABL001I12201; 2021-001286-20 (EudraCT Number)
Expanded Access: NCT04360005 (Available)
Record Dates: First submitted 2021-05-18; First posted 2021-06-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Myeloid Leukemia, Philadelphia Positive
Keywords: Asciminib; pediatric patients; Philadelphia chromosome positive chronic myeloid leukemia in chronic phase; Ph+ CML-CP; ABL001
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Asciminib (Experimental): This arm consists of 2 groups:
  * The pediatric formulation group where the dose is based on body weight (1.3mg/kg BID or 2.6 mg/kg QD)
  * The adult formulation group where participants will receive a flat dose of 40mg BID
  Interventions: Drug: Asciminib Pediatric formulation group; Drug: Asciminib Adult formulation group

INTERVENTIONS:
Drug: Asciminib Pediatric formulation group — Asciminib Pediatric formulation group: 1 mg film-coated granules in a size 0 capsule will be supplied, taken orally (capsules are a container for the granules and are not ingested):
  10 mg (10x 1 mg film-coated granules in capsule) 15 mg (15x 1 mg film-coated granules in capsule) 20 mg (20x 1 mg film-coated granules in capsule) 30 mg (30x 1 mg film-coated granules in capsule)
  Other Names: ABL001
Drug: Asciminib Adult formulation group — Asciminib Adult formulation group:
  40 mg tablets BID, taken orally. 20 mg tablets BID, taken orally.
  Other Names: ABL001

SUMMARY:
The aim of this study is to support development of asciminib in the pediatric population (1 to <18 years) previously treated with one or more TKIs. Full extrapolation of the efficacy of asciminib from adult to pediatric patients will be conducted. Full extrapolation is based on the concept that CML in the pediatric population has the same pathogenesis, similar clinical characteristics and progression pattern as in adults.

DETAILED DESCRIPTION:
The aim of this study is to support development of asciminib in the pediatric population (1 to <18 years) with Philadelphia chromosome positive chronic myeloid leukemia in chronic phase (PH+ CML-CP) previously treated with one or more Tyrosine kinase inhibitor (TKIs).

The primary objective of this study is to characterize the pharmacokinetic (PK) profile of asciminib in pediatric patients with the goal of identifying the pediatric formulation dose (fed) leading to asciminib exposure comparable to 40 mg BID in adult patients (fasted).

The pediatric formulation group will include at least 15 participants in each of the following two age categories: 1 to <12 years and 12 to <18 years; leading to at least 30 participants enrolled treated with the pediatric formulation. It will consist of a dose determination part (Part 1) and a cohort expansion (Part 2 BID regimen and Part 3 QD regimen).

In Part 1, 4-6 participants will be enrolled in order to obtain at least 4 participants evaluable for PK (these participants may be from either of the age categories described above). The initial starting dose will be based on body weight and will be administered BID with food.

Once the body weight adjusted dose has been determined in Part 1 of the study, the patients will be enrolled in Part 2 until at least 20 participants, including those who were included in Part 1, have been enrolled (10 per age group) in the pediatric formulation group. Once the interim safety and PK analysis 2 is completed for one of the age groups, the Part 3 QD regimen will open for the respective age group to enroll 10 patients (5 patients by age group).

Due to the fact that the pediatric formulation was in development and was not available, this study started with the recruitment of adolescent patients. These participants aged 14 to <18 years, weighing at least 40 kg receive the adult formulation at a flat dose of 40 mg BID under fasted conditions.

The total duration of the treatment period of the study will be 5 years (260 weeks). Participants who, according to Investigator's judgement, are benefiting from study treatment will remain on treatment up to the completion of the treatment period (Week 260/5 years). The primary analysis for the BID regimen is planned after all participants in Part 1 and 2 have completed at least 52 weeks of study treatment or discontinued earlier.

The primary analysis for combined regimen (BID+QD) is planned after all participants in Part 1, 2 and 3 have completed at least 52 weeks of study treatment or discontinued earlier.

ELIGIBILITY:
Inclusion Criteria:

- Male or female participants: Pediatric formulation group: ≥ 1 and less than 18 years of age at study entry. Adult formulation group: ≥ 14 and less than 18 years of age and body weight of ≥ 40 kg at study entry.

* Participants with Ph+ CML-CP must meet all of the following laboratory values at the screening visit. In the case where bone marrow blast and promyelocyte counts are available, these will be accepted if done within 56 days prior to the screening visit, to avoid unnecessary repetition of this test.

  1. < 15% blasts in peripheral blood and bone marrow
  2. < 30% combined blasts plus promyelocytes in peripheral blood and bone marrow
  3. < 20% basophils in the peripheral blood
  4. Neutrophils ≥ 1.5 x 10^9/L (or WBC ≥ 3 x 10^9/L if neutrophils are not available) and platelet count ≥ 100 x 10^9/L
  5. No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
* Prior treatment with a minimum of one TKI
* Failure (adapted from the 2020 European Leukemia Net (ELN) Guidelines Hochhaus et al 2020 and 2013 ELN Guidelines Baccarani et al 2013) or intolerance to the most recent TKI therapy at the time of screening.
* Performance status: Karnofsky ≥ 50% for patients ≥ 16 years of age, and Lansky ≥ 50 for patients < 16 years of age at the time of screening
* Participants must have adequate renal, hepatic, pancreatic and cardiac function
* Participants must have electrolyte values within normal limits or corrected to be within normal limits with supplements prior to first dose of study medication:
* Evidence of typical BCR-ABL1 transcript [e14a2 and/or e13a2] at the time of screening which are amenable to standardized RQ-PCR quantification.

Exclusion Criteria:

* Known presence of the T315I mutation prior to study entry or a BCR::ABL mutation with known resistance to study treatment any time prior to study entry.
* Known second chronic phase of CML after previous progression to AP/BC.
* Previous treatment with a hematopoietic stem-cell transplantation.
* Patient planning to undergo allogeneic hematopoietic stem cell transplantation.
* Cardiac or cardiac repolarization abnormality
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the Investigator could cause unacceptable safety risks or compromise compliance with the protocol
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
* History of acute or chronic liver disease.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug
* Pregnant or nursing (lactating) females.

Other protocol-defined inclusion/exclusion may apply.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary Pharmacokinetic (PK) parameter: AUClast | 52 weeks
  Goal: identifying the pediatric formulation dose (fed) leading to asciminib exposure comparable to 40 mg BID in adult patients (fasted).
Primary PK parameter: AUCtau | 52 weeks
  Goal: identifying the pediatric formulation dose (fed) leading to asciminib exposure comparable to 40 mg BID in adult patients (fasted).
Secondary PK parameter: Cmax | 52 weeks
  Goal: identifying the pediatric formulation dose (fed) leading to asciminib exposure comparable to 40 mg BID in adult patients (fasted).
Secondary PK parameter: Tmax | 52 weeks
  Goal: identifying the pediatric formulation dose (fed) leading to asciminib exposure comparable to 40 mg BID in adult patients (fasted).
Secondary PK parameter: Ctrough | 52 weeks
  Goal: identifying the pediatric formulation dose (fed) leading to asciminib exposure comparable to 40 mg BID in adult patients (fasted).

SECONDARY OUTCOMES:
Hematologic responses | 52 weeks
  Complete hematological response will be defined as all of the following present for ≥ 4 weeks:
  * WBC count < 10 x 10^9/L
  * Platelet count < 450 x 10^9/L
  * Basophils < 5%
  * No blasts and promyelocytes in peripheral blood
  * Myelocytes + metamyelocytes < 5% in peripheral blood
  * No evidence of extramedullary disease, including spleen and liver
Molecular responses | 52 weeks
  To assess pharmacodynamic markers of asciminib's anti-leukemic activity. Molecular response will be assessed by Breakpoint Cluster Region gene-Abelson proto-oncogene (BCR-ABL) 1 level.
Questionnaire on acceptability and palatability after first dose, 4 and 52 weeks | after first dose at Week 1 Day 1, 4 weeks, 52 weeks
  To assess acceptability and palatability of the pediatric formulation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- United States (8):
  - Indiana UH Riley H for CIU, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia University Medical Center New York Presbyterian, New York, New York
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Uni Of Texas MD Anderson Cancer Ctr, Houston, Texas
  - University Of Utah, Salt Lake City, Utah
- China (4):
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- France (4):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
- Germany (3):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Budapest, Hungary
- Italy (4):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Japan (3):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Wroclaw, Poland
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Seoul, South Korea
- Thailand (3):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Bursa, Nilufer

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com